CLINICAL TRIAL: NCT02153658
Title: A Prospective, Randomized, Open Label, Blinded Assessor, Trial Comparing Odor Levels Due to Different Hygiene Techniques When Using the PrePexTM Device
Brief Title: An Open Label, Blinded Assessor, Trial Comparing Odor Levels Due to Different Hygiene Methods With PrePexTM
Acronym: RMC-10
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Rwanda (Other Government)
Responsible Party: Principal Investigator, Vincent Mutabazi, Director of the Research Grants Unit, Ministry of Health, Rwanda
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Odor Study (RMC-10)
Record Dates: First submitted 2014-05-22; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Odor Levels of Study Arms
Keywords: PrePex; Odor; Cleaning technique; Male Circumcision; HIV; AIDS; Chlorhexidine; Soap
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (No Intervention): Subjects followed the current hygiene instructions, standard washing in a shower with soap.
- Arm 2 (Active Comparator): Subjects cleaned the foreskin with soapy water using a syringe once a day.
  Interventions: Procedure: Subjects cleaned the foreskin with soapy water using a syringe once a day.
- Arm 3 (Active Comparator): Subjects cleaned the foreskin with diluted chlorhexidine (1%) using a syringe once a day.
  Interventions: Procedure: Subjects cleaned the foreskin with diluted chlorhexidine (1%) using a syringe once a day.

INTERVENTIONS:
Procedure: Subjects cleaned the foreskin with soapy water using a syringe once a day.
  Arms: Arm 2
Procedure: Subjects cleaned the foreskin with diluted chlorhexidine (1%) using a syringe once a day.
  Arms: Arm 3

SUMMARY:
The PrePex is a WHO prequalified medical device for adult male circumcision for HIV prevention. The Government of Rwanda was the first country to implement the PrePex and acts as the leading Center of Excellence providing trainings and formal guidelines. As part of the Government's efforts to improve the PrePex implementation, it made efforts to improve the psychology acceptability of the PrePex by men and thus to increase the uptake with VMMC in sub-Saharan Africa.

Some men who gone through the PrePex procedure complained of foreskin odor while wearing the PrePex 3-7 days after it is placed. This complaint was identified as potential risk for the PrePex uptake. Researchers from Rwanda assumed there is a possible relation between the level of foreskin odor to the patient foreskin hygiene technique. It was speculated that a patient that follows an appropriate foreskin hygiene technique while wearing the device will have a significantly lower foreskin odor on day 7 than a patient who does not follow such technique. The Government of Rwanda decided to investigate those assumptions in a scientific way and conduct a study to test different hygiene cleaning methods in order to increase the acceptability of PrePex and mitigate the odor concern.

DETAILED DESCRIPTION:
Voluntary Medical Male Circumcision (VMMC) is a one-time, low cost intervention that shown to reduce men's risk of HIV infection by 53%-60% and by up to 73% in post-trial observation. Numerous papers on the topic have been published over the past two decades to elevate HIV prevention awareness, especially in sub-Saharan countries.

The World Health Organization (WHO) and the Joint United Nations Program on HIV/AIDS (UNAIDS) have endorsed innovative approaches to VMMC uptake in settings where HIV prevalence and incidence is high but male circumcision (MC) prevalence remains low in 14 target countries. Recent modelling commissioned by President's Emergency Plan For AIDS Relief (PEPFAR) and UNAIDS have agreed on an action plan to reach 80% coverage of VMMC in the 14 countries by 2015, this will entail performing roughly 20 million adult VMMC by 2015, averting approximately 3.36 million new HIV infections and saving US$16.5 billion.

The PrePex became the first medical device for adult male circumcision to receive WHO prequalification as an alternative to the conventional surgical circumcision methods already recognized by WHO. The PrePex VMMC procedure is bloodless and requires no injected anesthesia, suturing, or sterile setting, it applies controlled radial elastic pressure to the foreskin between a rigid Inner Ring and an Elastic Ring to cut off distal blood flow. After 7 days, the necrotic foreskin and the device are removed.

The Government of Rwanda was the first country to implement the PrePex and acts as the leading Center of Excellence providing trainings and formal guidelines. As part of the Government's efforts to improve the PrePex implementation, it made efforts to improve the psychology acceptability of the PrePex by men and thus to increase the uptake with VMMC in sub-Saharan Africa.

PrePex researchers from Rwanda have assumed that there is a possible relation between the level of odor from the foreskin to the foreskin hygiene technique. It was speculated that when a patient follows an appropriate foreskin hygiene technique while wearing the device, the odor before device removal (day 7) will be significantly lower than the odor of the foreskin of a subject who follows a less effective foreskin hygiene technique.

Providing scientific evidence of the direct relation between odor and specific foreskin hygiene technique, will allow VMMC implementing bodies to create a comprehensive and effective PrePex related hygiene guidelines and reduce the potential of complaints from men therefore, increasing the acceptability rate. A randomized, controlled, blinded study to assess the effectiveness of 3 different foreskin hygiene techniques was conducted at Rwanda Military Hospital Kigali, Rwanda during November 18th to December 4th, 2013.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  * Ages - 21 to 49 years
  * Subject wants to be circumcised
  * Uncircumcised
  * Able to understand the study procedures and requirements
  * Agrees to participate in one of the arms and to follow hygiene instructions
  * Agrees to have Independent blinded smell reviewers in the same room on Removal visit
  * Agrees that his partner will be interviewed via telephone
  * Agrees to abstain sexual intercourse for 6 weeks post device removal
  * Agrees to abstain from masturbation for 2 weeks post device removal
  * Agrees to return to the health care facility for follow-up visits (or as instructed) after his circumcision for a period of 1 week
  * Subject able to comprehend and freely give informed consent for participation in this study and is considered by the investigator to have good compliance for the study
  * Subject agrees to anonymous video and photographs of the procedure and follow up visits.

Exclusion Criteria:

* Active genital infection, anatomic abnormality or other condition, which in the opinion of the investigator prevents the subject from undergoing a circumcision
* Subject with the following diseases/conditions: phimosis, paraphimosis, warts under the prepuce, torn or tight frenulum, narrow prepuce, hypospadias, epispadias
* Known bleeding / coagulation abnormality, uncontrolled diabetes, by questionnaire
* Subject who have an abnormal penile anatomy or any penile diseases
* Subject that to the opinion of the investigator is not a good candidate
* Subject does not agree to anonymous video and photographs of the procedure and follow up visits.

Ages: 21 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in Dilution-to-Threshold" (D/T) values | Baseline, 3, 5 and 7 days
  The measurements were done by a Nasal Ranger device

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Mutabazi, M.D., Principal Investigator — RBC-Medical Research Centre (MRC); Jean Paul Bitega, M.D., Principal Investigator — Military Insurance Medical
Locations (1):
- Rwanda Military Hospital, Kigali, Rwanda

REFERENCES:
- [Derived] Mutabazi V, Bitega JP, Ngeruka LM, Karema C, Binagwaho A. Assessing Odor Level when Using PrePex for HIV Prevention: A Prospective, Randomized, Open Label, Blinded Assessor Trial to Improve Uptake of Male Circumcision. PLoS One. 2015 May 29;10(5):e0126664. doi: 10.1371/journal.pone.0126664. eCollection 2015. PMID 26023772
- See also: Biomedical Center — http://www.rbc.gov.rw/